CLINICAL TRIAL: NCT07049172
Title: Efficacy and Safety of Rituximab in Reducing Relapses in Children With Steroid-Sensitive Nephrotic Syndrome: An Open-label, Multi-center Clinical Study.
Brief Title: Rituximab and Targeted Nursing for Pediatric Nephrotic Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wuhan Children's Hospital (Other)
Responsible Party: Principal Investigator, Ting Xu, Principal investigator, Wuhan Children's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: WX19Q09
Record Dates: First submitted 2025-06-24; First posted 2025-07-03 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-06

CONDITIONS: Nephrotic Syndrome in Children
Keywords: rituximab; targeted nursing care; pediatric nephrotic syndrome; tacrolimus; steroid-dependent nephrotic syndrome; frequently relapsing nephrotic syndrome
MeSH Terms: conditions — Nephrotic Syndrome | interventions — Rituximab; Tacrolimus

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Rituximab with Targeted Nursing Care (Experimental): Patients received intravenous rituximab in conjunction with baseline glucocorticoid therapy and a standardized targeted nursing care program
  Interventions: Drug: Rituximab; Behavioral: Targeted Nursing Care; Drug: Baseline Glucocorticoid Therapy
- Tacrolimus with Targeted Nursing Care (Active Comparator): Patients received oral tacrolimus capsules in conjunction with baseline glucocorticoid therapy and a standardized targeted nursing care program identical to the study group.
  Interventions: Behavioral: Targeted Nursing Care; Drug: Baseline Glucocorticoid Therapy; Drug: Tacrolimus

INTERVENTIONS:
Drug: Rituximab — * Dosage: 375 mg/m²
  * Route: Intravenous infusion
  * Frequency: Once a week
  * Duration: 12 consecutive weeks
  * Details: Diluted in 5% glucose solution. Infusion started at 25 ml/h, increased by 25 ml/h every 30 minutes if no adverse reactions, up to 100-150 ml/h.
  Other Names: Rituxan®
  Arms: Rituximab with Targeted Nursing Care
Behavioral: Targeted Nursing Care — A structured, individualized nursing approach involving joint goal-setting. Included health education, psychological support, relaxation techniques, dietary care, lifestyle guidance, complication management, and medication guidance. Delivered throughout hospital stay and reinforced during monthly follow-ups.
Drug: Baseline Glucocorticoid Therapy — Patients already on maintenance glucocorticoids continued their regimen. For relapse at admission, IV methylprednisolone (2 mg/kg/day), then oral prednisone (2 mg/kg/day, max 60mg/day) tapered according to standard protocols.
Drug: Tacrolimus — * Dosage: Initial dose 0.05-0.1 mg/kg/day, adjusted to maintain target trough levels of 5-10 ng/mL.
  * Route: Oral
  * Frequency: Divided into two doses (morning and evening)
  * Duration: Throughout the 6-month study period.
  Other Names: Prograf®
  Arms: Tacrolimus with Targeted Nursing Care

SUMMARY:
This study investigated the combined impact of rituximab and targeted nursing care versus tacrolimus and targeted nursing care on efficacy, quality of life, adverse reactions, and recurrence rate in children with challenging (steroid-dependent or frequently relapsing) nephrotic syndrome. Ninety-one pediatric patients were randomized to either receive rituximab plus targeted nursing or tacrolimus plus targeted nursing, and outcomes were assessed over a 6-month period.

DETAILED DESCRIPTION:
Nephrotic syndrome in children, particularly steroid-dependent (SDNS) or frequently relapsing (FRNS) types, poses significant treatment challenges. While glucocorticoids are initial mainstays, second-line immunosuppressants like tacrolimus or rituximab are often required. Rituximab, a monoclonal antibody targeting CD20 on B-lymphocytes, has shown promise. Targeted nursing care, a patient-centered approach involving joint goal-setting and personalized interventions, aims to improve adherence and overall well-being. This study aimed to evaluate the synergistic effect of rituximab therapy combined with a structured targeted nursing care program compared to tacrolimus with the same targeted nursing care.

A total of 91 pediatric patients (aged 6-15 years) with SDNS or FRNS were enrolled from January 2021 to June 2023. They were randomized into a study group (n=46, rituximab + targeted nursing) and a control group (n=45, oral tacrolimus + targeted nursing). Both groups received baseline glucocorticoid therapy. The study group received intravenous rituximab (375 mg/m² weekly for 12 weeks). The control group received oral tacrolimus (0.05-0.1 mg/kg/day, adjusted to trough levels). Both groups received identical targeted nursing care protocols.

Outcomes compared included clinical efficacy (remission status), quality of life (IS-LQ questionnaire), incidence of adverse reactions, and recurrence rate over a 6-month follow-up. Peripheral blood CD19+ B-cell counts were monitored in the rituximab group. The study was approved by the institutional ethics committee, and informed consent was obtained.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of primary pediatric nephrotic syndrome, specifically steroid-dependent nephrotic syndrome (SDNS) or frequently relapsing nephrotic syndrome (FRNS), as defined by the Kidney Disease: Improving Global Outcomes (KDIGO) guidelines. (SDNS is defined as relapse occurring during tapering of glucocorticoids or within 14 days of discontinuation; FRNS is defined as ≥2 relapses within 6 months of initial response or ≥4 relapses in any 12-month period).
* Age between 6 and 15 years.
* Normal intellectual development and the ability to understand and communicate.
* Informed consent obtained from the guardians and assent from children capable of understanding.

Exclusion Criteria:

* Steroid-resistant nephrotic syndrome (SRNS).
* Severe renal insufficiency (according to KDIGO criteria or other relevant standards).
* Cognitive or mental disorders.
* Worsening condition upon admission necessitating intensive care.
* Parents unable to provide long-term care or unwilling to participate.
* Interruption of hospitalization for any reason.
* Prior treatment with rituximab or tacrolimus.
* Co-existing significant kidney, urinary system diseases (other than NS), or severe active urinary tract infection.
* Significant liver function impairment.
* Known hypersensitivity to rituximab or tacrolimus.

Ages: 6 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 91 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Total Effective Rate | At 6 months post-treatment initiation.
  The percentage of participants who achieved a "Significantly effective" or "Effective" response. Efficacy is defined based on remission status, renal function, and proteinuria levels. Total effective rate is calculated as the number of (Significantly effective + Effective) cases divided by the total number of cases in the group.
Recurrence Rate | Within the 6-month follow-up period after treatment initiation.
  Relapse defined as urinary protein ≥2+ or urinary protein quantity >50 mg/kg (or urine protein/creatinine ratio >2.0 mg/mg), occurring on three consecutive days within a 7-day period, after having achieved remission.

SECONDARY OUTCOMES:
Change in Quality of Life as Assessed by the Children's Subjective Quality of Life Questionnaire (IS-LQ) | Baseline and at 6 months post-treatment initiation.
  The IS-LQ consists of 60 items, scored from 1 to 4, with higher scores indicating better quality of life. Assesses six areas including cognitive, emotional, and overall functioning.
Adverse Reactions | During the 6-month study period.
  Any adverse reactions recorded, including infections, infusion reactions (for rituximab), hypertension, hyperglycemia, electrolyte disturbances, and gastrointestinal symptoms.

OTHER OUTCOMES:
Peripheral Blood CD19+ B-Cell Count | Monitored monthly in the study group during the 6-month follow-up.
  Absolute count of peripheral blood CD19+ B-cells, measured to confirm biological effect of rituximab (B-cell depletion, defined as CD19+ count <5 cells/μL or <1% of total lymphocytes). This measure applies to the Rituximab group only.

CONTACTS AND LOCATIONS:
Locations (1):
- Wuhan Children's Hospital, Wuhan, Hubei, China

REFERENCES:
- [Derived] He L, Mei H, Gu Y, Liu Z, Yang L, Li X, Wang X, Xu T. Combined impact of rituximab and target care on efficacy, quality of life, adverse reactions and recurrence rate in children with nephrotic syndrome: a randomized controlled trial. BMC Pediatr. 2025 Sep 24;25(1):691. doi: 10.1186/s12887-025-06070-0. PMID 40993587